CLINICAL TRIAL: NCT03951415
Title: Durvalumab and Olaparib in Metastatic or Recurrent Endometrial Cancer
Acronym: DOMEC
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Leiden University Medical Center (Other)
Collaborators: Amsterdam University Medical Center (Other); Erasmus Medical Center (Other); Maastricht University Medical Center (Other); The Netherlands Cancer Institute (Other); Radboud University Medical Center (Other); University Medical Center Groningen (Other); UMC Utrecht (Other); AstraZeneca (Industry)
Responsible Party: Principal Investigator, J.R. Kroep, Principal Investigator, Leiden University Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DOMEC
Record Dates: First submitted 2019-04-30; First posted 2019-05-15 (Actual); Last update posted 2021-04-01 (Actual); Status verified 2021-03

CONDITIONS: Endometrial Neoplasms; Uterine Neoplasms; Endometrium Cancer
Keywords: Poly (ADP-ribose) Polymerase Inhibitors; Antibodies, Monoclonal; Checkpoint Inhibitors; olaparib; durvalumab; Anti-PD-L1
MeSH Terms: conditions — Endometrial Neoplasms; Uterine Neoplasms | interventions — Poly(ADP-ribose) Polymerase Inhibitors; olaparib; durvalumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- PARP inhibitor and Anti-PD-L1 (Experimental): olaparib tablets 300mg twice daily orally and durvalumab 1500mg by IV infusion every 4 weeks
  Interventions: Drug: PARP inhibitor and Anti-PD-L1

INTERVENTIONS:
Drug: PARP inhibitor and Anti-PD-L1 — olaparib tablets 300mg twice daily orally and durvalumab 1500mg by IV infusion every 4 weeks
  Other Names: olaparib; durvalumab; PARP inhibitor; Anti-PD-L1 Monoclonal Antibody

SUMMARY:
The DOMEC trial is designed as a Dutch Gynecological Oncology Group (DGOG), prospective, multi-center, phase II study for 55 patients with advanced (recurrent, refractory or metastatic) endometrial cancer or carcinosarcoma of the uterus to investigate the efficacy of the combination therapy of olaparib tablets and durvalumab IV.

DETAILED DESCRIPTION:
The prognosis of recurrent or persistent endometrial carcinoma not amenable to local therapy is poor. First line therapy exists of platinum-based chemotherapy or hormonal therapy. No standard subsequent-line therapy has been described.The combination of Poly(ADP-ribose) polymerases (PARP) inhibition and Programmed death-ligand 1 (PD-L1) blocking has great potential in the treatment of recurrent endometrial cancer. The DOMEC trial is designed to investigate this treatment combination among all molecular subgroups.

The DOMEC trial is designed as a DGOG, prospective, multi-center, phase II study for 55 patients with advanced (recurrent, refractory or metastatic) endometrial cancer, including carcinosarcoma of the uterus. Patients must have had one prior platinum-based chemotherapeutic regimen or not be able/willing to get chemotherapy. The aim is to investigate the efficacy of the combination therapy of olaparib tablets 300mg twice daily orally and durvalumab 1500mg by IV infusion every 4 weeks in terms of progression free survival. Secondary objectives are to investigate objective response rate, overall survival, safety and predictive biomarkers.

ELIGIBILITY:
Inclusion criteria:

* Written informed consent
* Age > 18 years old
* Histologically confirmed diagnosis of endometrial cancer or carcinosarcoma of the endometrium.
* Metastatic disease or locally advanced tumor not amenable to local therapy.
* Documented progressive disease before enrolment.
* Measurable lesions outside irradiated field or progressive measurable lesions in irradiated area
* Not eligible for hormonal therapy (because of negative hormone receptor/poor differentiation, or after failure of hormonal therapy).
* Previous failure of chemotherapy, or refusal to undergo chemotherapy or chemo-naive patients not suitable for chemotherapy.
* WHO performance 0-1
* Adequate organ system function as measured within 28 days prior to administration of study treatment, as defined below:

  * Haemoglobin ≥ 10.0 g/dL, with no blood transfusion in the past 28 days.
  * Absolute neutrophil count (ANC) ≥ 1.5 x 109/L
  * Platelet count ≥ 100 x 109/L
  * Total bilirubin ≤ 1.5 x institutional upper limit of normal (ULN) (not applicable to Gilbert's syndrome)
  * Aspartate aminotransferase (AST) (Serum Glutamic Oxaloacetic Transaminase (SGOT)) / Alanine aminotransferase (ALT) (Serum Glutamic Pyruvate Transaminase (SGPT)) ≤ 2.5 x ULN unless liver metastases are present in which case they must be ≤ 5x ULN
  * Patients must have creatinine clearance estimated of ≥51 mL/min estimated using the Cockcroft-Gault equation or 24 hr urine clearance.
* Life expectancy of at least 16 weeks.
* Measurable disease as defined by RECIST 1.1 criteria
* Able to swallow and retain oral medication.
* A female is eligible to enter and participate in this study if there is:

Exclusion criteria:

* Participation in another clinical study with an investigational product during the last month or previous enrolment in the present study.
* Any previous treatment with PARP inhibitor, including olaparib and/or any previous treatment with a PD1 or PD-L1 inhibitor
* History of another primary malignancy except for malignancy treated with curative intent and with no known active disease ≥5 years before the first dose of investigational product and of low potential risk for recurrence or adequately treated non-melanoma skin cancer, lentigo maligna or carcinoma in situ.
* History of leptomeningeal carcinomatosis, symptomatic uncontrolled brain metastases (≤2mg/ day corticosteroids started ≥4 weeks prior to treatment is accepted) and spinal cord compression (unless received definitive treatment and clinically stable for 28 days) .
* Resting ECG with QTc > 470 msec on 2 or more time points within a 24 hour period or family history of long QT syndrome
* Concomitant use of known strong or moderate CYP3A inhibitors and inducers.
* Any unresolved toxicity NCI CTCAE Grade ≥2 from previous anticancer therapy with the exception of alopecia, vitiligo, and the laboratory values defined in the inclusion criteria.
* Current or prior use of immunosuppressive medication within 14 days before the first dose of durvalumab (except intranasal and inhaled corticosteroids or systemic prednisone ≤ 10 mg/day)
* Major surgery ≤2 weeks of starting study treatment
* History of active primary immunodeficiency
* Active or prior documented autoimmune or inflammatory disorders, with exception of: vitiligo or alopecia, hypothyroidism stable on hormone replacement, any chronic skin condition that does not require systemic therapy, celiac disease controlled by diet alone
* Patients unable to swallow orally administered medication and patients with gastrointestinal disorders likely to interfere with absorption of the study medication.
* Active infection including tuberculosis, hepatitis B/C and HIV
* Patients with an expected or known hypersensitivity to olaparib or durvalumab or any of the excipients of the products.
* Previous allogenic bone marrow transplant or double umbilical cord blood transplantation (dUCBT).
* Receipt of live attenuated vaccine within 30 days prior to the first dose of IP.
* Pregnancy or breastfeeding

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 55 (Actual)
Dates: Start 2019-07-08 (Actual); Primary Completion 2021-08-01 (Estimated); Study Completion 2021-08-01 (Estimated)

PRIMARY OUTCOMES:
Progression free survival (PFS) | 6 months
  PFS will be counted from the date of registration until the first observation of radiological progressive disease according to RECIST 1.1 criteria or death due to any cause, whichever occurred first.

SECONDARY OUTCOMES:
Objective response rate (ORR) | 12 weeks
  according to RECIST 1.1 criteria
Overall survival (OS) | Through study completion, up to 36 months
  OS will be determined from the date of registration until death from any cause.
Adverse events | Through study completion, up to 36 months
  Assessed by NCI Common Terminology Criteria for adverse Events (CTCAE) version 5.0
Predictive biomarkers in tumor biopsy | At baseline
  MMRd/POLE, HR status, quantification of CD3,CD4,CD8,CD103,CD161,PD-1,LAG3,CTLA-4,NKG2A,GOXp3 positieve T cells, NK cells, percentage PD-L1 on myeloid cells/tumorcells, quantification of myeloid cell infiltration (CD68,CD14,CD33,CD163) in tumor biopsies.

OTHER OUTCOMES:
Functional HRD assay (optional) | At baseline
  Extra biopsy
Immunological effects of PARP-1 inhibition (optional) | Change From Baseline to 6 weeks and 12 weeks
  Tests for T cell and APC functionality measured by the measurement of recall antigen responses and mixed lymphocyte cultures, respectively, the levels of regulatory T cells, activation markers on T cells and DC).
Predictive biomarkers for PD-L1 blocking in blood (optional) | Change From Baseline to 6 weeks and 12 weeks
  e.g. monocyticMDSC levels, DC levels, inhibitory marker expression, neutrophil-to-lymphocyte ratio, absolute lymphocyte count, T-cell reactivity during PD-L1 blocking, T-cell cytokine expression after SEB activation

CONTACTS AND LOCATIONS:
Locations (8):
- Netherlands (8):
  - Amsterdam UMC, AMC, Amsterdam
  - NKI-AVL, Amsterdam
  - Universitair Medisch Centrum Groningen, Groningen
  - Leiden University Medical Center, Leiden
  - Academisch Ziekenhuis Maastricht, Maastricht
  - RadboudMC, Nijmegen
  - Erasmus MC, Rotterdam
  - Universitair Medisch Centrum Utrecht, Utrecht

IPD SHARING:
Plan to Share IPD: No